CLINICAL TRIAL: NCT01335425
Title: The Rolandic Epilepsy/ESES/Landau-Kleffner Syndrome and Correlation With Language Impairment Study
Acronym: REL
Status: Completed | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Epilepsiecentrum Kempenhaeghe (Industry)
Responsible Party: Principal Investigator, René Besseling, M Sc, Maastricht University Medical Center
Other Study IDs: 10-3-044; NCT01248559 (obsolete NCT alias)
Record Dates: First submitted 2011-04-13; First posted 2011-04-14 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-09

CONDITIONS: Rolandic Epilepsy; Nocturnal Frontal Lobe Epilepsy; Landau-Kleffner Syndrome; Electrical Status Epilepticus During Slow Wave Sleep
Keywords: Language problems; childhood epilepsy; bening (rolandic) epilepsy (of childhood) with centro temporal spikes; brain maturation; structral connectivity; functional connectivity
MeSH Terms: conditions — Epilepsy, Rolandic; Landau-Kleffner Syndrome; Epilepsy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
In clinical practice language impairment is frequently reported in association with nocturnal epileptiform activity. There is a spectrum of epileptic conditions that are characterized by nocturnal epileptiform activity. From mild to severe this spectrum involves: Rolandic epilepsy (RE), nocturnal frontal lobe epilepsy (NFLE), Landau-Kleffner syndrome (LKS) and electrical status epilepticus during slow wave sleep (ESES). The exact characteristic of the relationship between nocturnal epileptiform activity and language impairment is yet to be explored. The investigators suggest that nocturnal epileptiform EEG discharges and nocturnal epileptic seizures during development will cause diseased neuronal networks that involve language. The diseased neuronal networks are less efficient compared with normal neuronal networks.

Objective: Identification of a diseased neuronal network characteristic in children with nocturnal epileptiform activity, which can explain language impairment in these children. For this the investigators will use functional magnetic resonance imaging (MRI) to analyse brain activity and diffusion weighted MRI to investigate white matter connectivity.

ELIGIBILITY:
Inclusion Criteria:

* aged between 6-18
* diagnosis of Rolandic epilepsy (or other childhood epilepsies as listed in study population description)

Exclusion Criteria:

* structural brain lesions which might influence cognition

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children aged 6 to 18 years seen in tertiary referral center for epilepsy Kempenhaeghe with a proven diagnosis of Rolandic epilepsy and without intracerebral lesions (e.g. tumour) on structural MRI or other pathology, which may influence cognition.
  In addition, children with electrical status epilepticus of sleep (ESES), ESES-like, or Landau-Klefner syndrome might be included.
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2010-10; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Mechanism that causes language problems in childhood epilepsy | course of study
  Morphological, anatomical or functional correlate that can explain the comorbidity of language problems in childhood epilepsy. In Rolandic epilepsy, e.g., the epileptic focus is in the brain motor strip, and from classical anatomy no connection is known from the motor strip to the language areas. Think of deviations in the brain such as cortical thinning in both regions or aberrant functional or anatomical networks linking both regions.

CONTACTS AND LOCATIONS:
Locations (1):
- Epilepsiecentrum Kempenhaeghe, Heeze, North Brabant, Netherlands